CLINICAL TRIAL: NCT01647776
Title: Screening and Risk Factors of Colon Neoplasia
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE1207; SPORE 2 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2012-07-05; First posted 2012-07-24 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Colon Cancer
Keywords: Colon Neoplasia; Colorectal carcinoma; colon cancer; colon polyp; colonoscopy; sDNA test; FIT tests (fecal immunochemical test); relating colon neoplasia to obesity, type 2 diabetes; colonoscopy and pathology confirmed advanced adenomas
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Colonic Polyps; Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Urine, Stool samples, Colon polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals without colon polyps
  Interventions: Other: Stool DNA Test; Procedure: biopsies of rectal and colon mucosa; Other: Questionnaires
- Individuals with colon polyps
  Interventions: Other: Stool DNA Test; Procedure: biopsies of rectal and colon mucosa; Other: Questionnaires

INTERVENTIONS:
Other: Stool DNA Test — Stool DNA test is done prior to the colonoscopy.
  Other Names: sDNA
Procedure: biopsies of rectal and colon mucosa — During the standard of care colonoscopy biopsies of rectal and colon mucosa will be taken for analysis of 15-PGDH pathway factors [levels of prostaglandin E2 (PG E2), and mRNA for 15-PGDH, COX-1 and COX-2 expression] as markers of risk of developing adenoma.
Other: Questionnaires — A Food Frequency Questionnaire (FFQ), a Meat Preparation Questionnaire (MPQ), and a Physical Activity Questionnaire (PAQ), all developed at the University of Arizona Cancer Center will be used to collect dietary and physical activity data. Risk Factor Questionnaire (RFQ) developed by the University of Southern California will be used to collect general risk information. Stool (sDNA) test patient satisfaction survey.
  Other Names: Food Frequency Questionnaire (FFQ); Meat Preparation Questionnaire (MPQ); Physical Activity Questionnaire (PAQ); Risk Factor Questionnaire (RFQ)

SUMMARY:
The investigators propose a screening population-based study to systematically evaluate the accuracy and clinical relevance of sDNA testing as a potential alternative to colonoscopy screening. In addition, the investigators propose a genetic epidemiologic study of the relation between colon polyps, an established precursor of colon cancer, and two factors that may influence risk for colon cancer: candidate genes and diet.

DETAILED DESCRIPTION:
Colorectal carcinoma is currently the second most common fatal cancer in the United States, and is largely preventable through the use of screening in the asymptomatic population. Although colonoscopy is considered to be the most accurate 'gold standard' screening test, there are a significant proportion of eligible patients who decline colonoscopy or in whom colonoscopy is not readily available. More recently, testing for aberrant molecular/genetic markers in stool DNA (sDNA) is emerging as a promising alternative to colonoscopy, and some professional society guidelines have endorsed the use of sDNA testing in the early detection of colorectal cancer. However, despite some guidelines that endorse sDNA testing primarily for the detection of colorectal cancer, data on the efficacy of sDNA testing for advanced adenomas, and hence prevention of colorectal cancer, are limited.

Colon carcinogenesis is a multifactorial and multistep process that involves both genetic and environmental influences. Diet clearly plays an important role. However, despite extensive research, there has been limited success in identifying such specific dietary and nutritional factors. In particular, a number of within-population studies, including several randomized trials, have yielded conflicting results and cast serious doubt on the hypothesized central role of dietary fat and fiber in colon carcinogenesis. In contrast, there is increasing evidence relating colon neoplasia to obesity, type 2 diabetes and related metabolic abnormalities. These results, together with the marked and consistent similarities in the dietary and lifestyle risk factors for type 2 diabetes and colon neoplasia have led to the notion that insulin resistance resulting from energy imbalance (excess energy intake, physical inactivity, and obesity) may be the underlying link between these two entities. Indeed, the insulin resistance-colon neoplasia hypothesis could account for many of the dietary and lifestyle risk factors of colon neoplasia and for its high incidence in Western countries. The fact that the incidences of obesity, insulin resistance syndrome, and type 2 diabetes are escalating at epidemic pace in the Western societies makes the exploration of the insulin resistance-colon neoplasia hypothesis a subject of pressing priority.

A Food Frequency Questionnaire (FFQ), a Meat Preparation Questionnaire (MPQ), and a Physical Activity Questionnaire (PAQ), all developed at the University of Arizona Cancer Center will be used to collect dietary and physical activity data.The FFQ, MPQ and PAQ questionnaires will be self-administered by each subject according to detailed written instructions, and they are mailed to the participant with the consent forms. Subjects will be asked to donate whole blood and urine samples on the day of routine colonoscopy exams. These samples will be looked at for disease markers. Stool samples will be collected to evaluate its use at detecting colon polyps using the sDNA Test and 2 FIT tests (fecal immunochemical test).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing routine colonoscopy at University Hospitals, Cleveland Ohio

Exclusion Criteria:

* Unable to give written consents
* Unable to fill the questionnaires
* A history of polyps within the past 10 years (except hyperplastic polyps)
* Family history of Familial Adenomatous Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC)
* Personal history of inflammatory bowel disease
* Personal diagnosis of any cancer, with the exception of non-melanoma skin cancer
* Any major colon surgeries (e.g. resectioning)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Average-risk patients undergoing colonoscopy at screening endoscopy centers in the University Hospitals of Cleveland system.
Sampling Method: Probability Sample
Enrollment: 3315 (Actual)
Dates: Start 2012-04-01; Primary Completion 2015-08-11 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Stool DNA (sDNA) Feasibility and Compliance | within 12 weeks prior to the colonoscopy
  For this aim, we will recruit a sub-sample of the study participants to perform the sDNA test for aberrantly methylated markers in addition to their colonoscopy to assess willingness to participate, compliance with test protocol and patient satisfaction to determine potential for a larger study to evaluate the effectiveness of this test for detection of colon adenomas.
Efficacy of sDNA testing for the detection of advanced adenomas | prior to the colonoscopy
  For the sDNA test aims, the primary goals are to assess the sensitivity and specificity of sDNA testing for the detection of advanced adenomas, and to compare the performance of the Exact sDNA Panel with that of FIT. The sensitivity and specificity of sDNA and FIT will be estimated based on the concordance and discordance of advanced adenomas detected against that of colonoscopy as the gold standard

SECONDARY OUTCOMES:
Concordance/discordance between tissue and stool DNA aberrant methylation markers | Stool sample within 2 weeks of colonoscopy
  Biopsies of rectal and colon mucosa collected at the beginning of the colonoscopy for analysis of 15-PGDH pathway factors [levels of prostaglandin E2 (PG E2), and mRNA for 15-PGDH, COX-1 and COX-2 expression] as markers of risk of developing adenoma.
Persistence of positive sDNA testing after removal of advanced adenomas | at 12 months after initial colonoscopy
  For this aim we will follow-up participants who have had positive sDNA tests and at least one advanced adenoma removed during colonoscopy. At 12 months after their initial sDNA test and colonoscopy, we will ask them to repeat the sDNA test in addition to colonoscopy recommended by their physician as standard of care.
Assess the frequency of missed or occult colonic and upper gastrointestinal neoplasia in patients with initially normal colonoscopies and persistently positive sDNA testing. | at 12 months after initial colonoscopy
  For this aim we will follow-up participants who have had positive sDNA tests and negative colonoscopy (i.e., no adenomatous polyps observed at initial colonoscopy). At 12 months after their initial sDNA test and colonoscopy, we will ask them to repeat the sDNA test. If this second sDNA test is also positive, the participant will be offered the opportunity to have both a colonoscopy and an upper GI endoscopy (also called esophagogastroduodenoscopy or EGD)
Insulin Resistance Syndrome | at the time of the colonoscopy
  Use latent structural equation models to fully incorporate information on the overall relations among insulin resistance syndrome pathway factors and colon polyps, including both direct and indirect effects as well as interactions between these factors.
Analyses stratified by ethnicity (Caucasians versus African Americans), and gender. | at the time of the colonoscopy
  The analysis by ethnicity is of particular interest in sDNA testing as there is evidence that large right-sided adenomas are more prevalent among African Americans, and this ethnic population is less likely to receive screening colonoscopy as compared to Caucasians. Furthermore, the ability of sDNA and FIT for the detection of nonadvanced adenomas will be evaluated. These lesions will be defined as adenomas that are less than 1 cm in diameter and without evidence of high grade dysplasia.
Examine the impact of candidate gene variants in the insulin-GH-IGF-IRS axis on colon polyps. | at the time of the colonoscopy
  Evaluate whether each of the following candidate gene polymorphisms and their haplotypes are linked to colon polyps: 1) Insulin; 2) Growth Hormone; 3) IGF-1; and 4) IRS-1.
Evaluate the association of dietary patterns, glycemic index (GI) and glycemic load (GL) with colon polyps. | at 12 months
  Conceptually, dietary patterns represent a broader picture of human diet, and thus may be more predictive of disease risk than individual foods or nutrients. In addition, there is growing evidence relating GI and/or GL to risks of obesity, type 2 diabetes as well as colon neoplasia. Therefore, we hypothesize that high dietary GL and/or GI, and/or a Western dietary pattern defined by a diverse array of dietary factors are associated with increased risk of colon polyps.
Synthesize the information on candidate genes and diet by looking at their joint effects on colon polyps | at the time of the colonoscopy
  1) investigate their potential joint actions [i.e., gene-diet and gene-gene]; 2) use a latent structural equation modeling approach to comprehensively evaluate these factors' potential direct as well as indirect (mediated by insulin resistance syndrome) impact, on colon polyps.
To investigate the association of activated (phosphorylated) IRS1, AKT and mTOR with colon adenomas. | at the time of the colonoscopy
  We will compare the immunohistochemistry of phosphorylated IRS1, AKT and mTOR in colon adenoma tissues with that in colon tissues from healthy control patients. Investigate the effect of obesity on the activation of the IRS1, AKT and mTOR by stratifying our cases and controls into lean and obese individuals. Evaluate the effects of serum levels of insulin, glucose, and insulin resistance index (HOMA-IR) on the activation of the IRS1, AKT and mTOR in colonic tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Willis, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States